CLINICAL TRIAL: NCT06043557
Title: Patient Satisfaction and Reflection on Drain Placement in Abdominoplasty and Panniculectomy
Brief Title: Patient Satisfaction and Reflection on Drain Placement
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00100958
Record Dates: First submitted 2023-09-12; First posted 2023-09-21 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Abdominoplasty; Panniculectomy
Keywords: Abdominoplasty; plastic surgery; panniculectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- left side lateral and right side medial (Active Comparator): left side lateral and right side medial
  Interventions: Procedure: Drain Placement
- right side lateral with left side medial (Active Comparator): right side lateral with left side medial
  Interventions: Procedure: Drain Placement

INTERVENTIONS:
Procedure: Drain Placement — Surgical placement of drain based on subject randomization.

SUMMARY:
The purpose of this research study is to evaluate the ideal drain placement in patients undergoing abdominoplasty or panniculectomy. There are currently no patient reported outcome measurements on ideal drain placement and this study aims to collect objective and patient reported measures to standardize ideal drain placement.

In this study a medially and laterally placed drain will be compared to each other in each study participant. In this study subject will have two drains. One will be lateral and one medial. The drains will be secured and dressed in the same manner. At subjects planned post-operative visits, subjects will be asked to complete surveys to evaluate their experience with the drains. This study will not require additional clinic visits for study purposes.

DETAILED DESCRIPTION:
The primary goal of this proposal is to assess patient perspectives and satisfaction with the location of their drains after abdominoplasty and/or panniculectomy. This will be conducted as a prospective observational trial, where patients with scheduled abdominoplasty and/or panniculectomy will be invited to participate. Patients will be randomized to either A) left side lateral and right side medial or B) right side lateral with left side medial. Randomization will occur before study initiation with group A or group B being assigned to a study enrollment number.

ELIGIBILITY:
Inclusion Criteria:

* age 18 or older
* patient of Department of Plastic and Reconstructive Surgery
* able to sign English language Consent form
* undergoing either abdominoplasty and/or panniculectomy.

Exclusion Criteria:

* Patients with unilateral drain placement, unable to sign English language consent form
* Patient under the age of 18.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Patient preference of surgical drain placement | 1 week post surgery
  Patients will complete a survey about their experience with the pertinent securement method/drain site - questions are essay style without a score or range
  In the survey we created the level of negative factors (pulling, tugging, pain) as well as positive (ease of drain care, ease of personal hygiene) will be on a 1-100 scale. Therefore each side will get a conglomerate score of the following:
  Total score = positive scores (average) - negative scores (average)
  This result will be tabulated for each patient and used as a group analysis for preference. (Average scores for each side from all patients compared to one another.)

SECONDARY OUTCOMES:
Number of days until drain removed | day of surgery up to 10 days
  tracking number of days

CONTACTS AND LOCATIONS:
Overall Officials: Adam Katz, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No